CLINICAL TRIAL: NCT04479514
Title: Preventative Skin Care for Children Undergoing Targeted CNS Tumor Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Jennifer Huang, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-579
Record Dates: First submitted 2020-07-15; First posted 2020-07-21 (Actual); Results first posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Pediatric Cancer; CNS Tumor, Childhood; Skin Inflammation
Keywords: Pediatric Cancer; CNS Tumor, Childhood; Skin Inflammation
MeSH Terms: conditions — Neoplasms; Central Nervous System Neoplasms; Dermatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Preventative Skin Care Routine (Experimental): Participants will perform a preventative skin care routine that includes daily sun protection, daily gentle skin care and every-other-day dilute bleach baths for the duration of the study.
  Participants will receive skin examinations and complete a survey about their skin condition at the initial visit when anti-cancer treatment is started, at six weeks after the start of treatment, and at twelve weeks after the start of treatment.
  Interventions: Other: Warm Baths or Showers; Other: Moisturizer; Drug: SPF 30 or Higher Suncreen; Other: Sun Protective Clothing; Behavioral: Limited Sun Exposure; Other: Dilute bleach baths

INTERVENTIONS:
Other: Warm Baths or Showers — Daily warm baths or showers
Other: Moisturizer — moisturizers applied daily immediately after bathing
Drug: SPF 30 or Higher Suncreen — Mineral based sunscreen of SPF 30 or higher applied on a daily basis on all sun exposed areas.
  Other Names: i.e. Neutrogena, Aveeno, Cerave, Blue Lizard
Other: Sun Protective Clothing — Sun protective clothing worn when outdoors
Behavioral: Limited Sun Exposure — Limit sun exposure during peak hours of 10am-4pm
Other: Dilute bleach baths — Warm 10-15 minute dilute bleach baths every other day

SUMMARY:
This research study is examining a preventive skin care regimen for children diagnosed with a brain tumor and receiving anti-cancer therapy with a MEK, Pan-RAF, or BRAF inhibitor.

DETAILED DESCRIPTION:
This prospective, single-arm phase 2 clinical trial is looking at whether gentle skin care, sun protection and dilute bleach baths might decrease the chances or the severity of skin changes that occur during treatment for brain tumors.

The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.

Participants will receive a study treatment regimen that involves a daily sun protection, daily gentle skin care and every-other-day dilute bleach baths for the duration of the study.

Participants enrolled in this study, will be in this research study during the course of their anti-cancer treatment and receive skin examinations and complete a survey about their skin condition at the initial visit when anti-cancer treatment is started, at six weeks after the start of anti-cancer treatment, and at twelve weeks after the start of anti-cancer treatment.

Participants will be followed for twelve weeks.

It is expected that about 20 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with a brain tumor between ages 6 months old -18 years old and will undergo treatment with at least one of the following:

  1. Targeted BRAF inhibitor therapy to treat the brain tumor
  2. Targeted MEK inhibitor therapy to treat the brain tumor
  3. Targeted pan-RAF inhibitor therapy to treat the brain tumor
* Subjects may participate in other studies, including therapeutic trials.
* Ability to comply with PSCR including sun protection, gentle skin care and every other day dilute bleach baths.
* Ability to understand and/or the willingness of their parent or legally authorized representative to sign a written informed consent document.

Exclusion Criteria:

* Diagnosed with brain tumor at > 18 years old
* No data in medical records regarding treatment exposures
* Treated with a BRAF, MEK or pan-RAF inhibitor in the last three months
* Past or present allergic reaction to bleach
* Past or present allergic reactions to sunscreen and/or creams, lotions, emollients to be utilized in this study

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2025-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Huang, MD, Principal Investigator — Boston Children's Hospital
Locations (2):
- United States (2):
  - Boston Children's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Preventative Skin Care Routine: Participants will perform a preventative skin care routine that includes daily sun protection, daily gentle skin care and every-other-day dilute bleach baths for the duration of the study.
  Participants will receive skin examinations and complete a survey about their skin condition at the initial visit when anti-cancer treatment is started, at six weeks after the start of treatment, and at twelve weeks after the start of treatment.
  Warm Baths or Showers: Daily warm baths or showers
  Moisturizer: moisturizers applied daily immediately after bathing
  SPF 30 or Higher Suncreen: Mineral based sunscreen of SPF 30 or higher applied on a daily basis on all sun exposed areas.
  Sun Protective Clothing: Sun protective clothing worn when outdoors
  Limited Sun Exposure: Limit sun exposure during peak hours of 10am-4pm
  Dilute bleach baths: Warm 10-15 minute dilute bleach baths every other day
Period: Overall Study
Arm/Group | Preventative Skin Care Routine
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Preventative Skin Care Routine
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 10.6 [4.5 to 20.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 10
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 7
  Canada | 7

OUTCOME MEASURES:

1. Primary Outcome: Rate of Cutaneous Reaction
Description: Proportion (percentage) of patients with one or more cutaneous reaction to targeted BRAF, MEK, or Pan-RAF inhibitor therapy
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Preventative Skin Care Routine
Number analyzed (Participants) | 14
Participants | 7

2. Secondary Outcome: Overall Cutaneous Reaction Severity
Description: Measured by the Common Terminology Criteria for Adverse Events (CTCAE)
Time Frame: 12 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Xerosis Severity
Description: Measured by the Overall Dry Skin Score (ODS)
Time Frame: 12 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Hand Foot Syndrome Severity
Description: Measured by the Hand-Foot Skin Reaction and Quality of Life Score (HFS-14)
Time Frame: 12 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Pediatric Quality of Life
Description: Pediatric Quality of Life Inventory (PedsQL)
Time Frame: 12 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Children's Dermatology Quality of Life
Description: Children's Dermatology Life Quality Index (CDLQI)
Time Frame: 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 week period
Arm/Group | Preventative Skin Care Routine
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-24): https://cdn.clinicaltrials.gov/large-docs/14/NCT04479514/Prot_SAP_000.pdf
  • Informed Consent Form (2021-12-10): https://cdn.clinicaltrials.gov/large-docs/14/NCT04479514/ICF_001.pdf